CLINICAL TRIAL: NCT06466330
Title: Efficacy of Microparticle Geniculate Artery Embolization in Total Knee Prosthesis Patients With Pain Resistant to Medical Treatment. A Prospective Randomized Controlled Trial
Acronym: EPROGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Societe Francaise de Rhumatologie (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EPROGE
Record Dates: First submitted 2024-06-10; First posted 2024-06-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Knee Pain Chronic; Knee Pain Swelling
Keywords: total hip replacement; pain
MeSH Terms: conditions — Pain | interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the interventional radiologist cannot be blinded, given the procedure (embolization with microparticles) . This means that the patient and the principal investigator at each center involved in the clinical evaluation of the patient will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization (Experimental): The genicular artery embolisation procedure identifies abnormal blood vessels in the knee via angiography. Through groin access and puncture of the femoral artery through a microcatheter, microspheres (Embozene) will be injected into this area.
  Interventions: Device: microparticles; Procedure: embolization
- Placebo (Sham Comparator): In the control (sham) arm patients will undergo angiography but there will be injection of saline.
  Interventions: Procedure: sham embolization

INTERVENTIONS:
Device: microparticles — inert microparticles
  Arms: Embolization
Procedure: embolization — Injection of inert microparticles in neovessels using a microcatheter
  Arms: Embolization
Procedure: sham embolization — injection of saline solution
  Arms: Placebo

SUMMARY:
The goal of this clinical investigation is to evaluate the effectiveness on pain of arterial occlusion (embolization) of neovessels by microparticle in a double-blind sham controlled randomised trial in patients with persistent pain on a total knee prosthesis (TKP), inserted for gonarthrosis, despite well-conducted medical treatment. The study patient population will consist of up to 112 subjects with knee pain for at least 3 months that is resistant to conservative treatment measures. Subjects will be treated with knee embolisation or saline in the sham arm. The efficacy of embolization will be judged on the basis of the following criteria: improvement in pain, mobility, use of pain medication, adverse effects of embolization and duration of improvement.

After verification of eligibility criteria, patients with painful total knee prosthesis will be randomized to either the embolization group or the control group. Embolization will be performed using microparticles (Embozene® Microspheres 100 microns from Varian), for the treatment group. For the "sham " group, only diagnostic arteriography will be performed without injection of microparticles. Subjects will be followed up at 1, 3, 6 and 12 months.

DETAILED DESCRIPTION:
Rational: One hundred thousand total knee replacements (TKRs) are fitted annually in France. Twenty percent of patients who have undergone a TKR have residual pain unrelated to a technical fault or loosening. This pain is a major handicap in everyday life, with no effective therapeutic solution. Arterial embolization for therapeutic purposes is rapidly gaining ground in a variety of pathologies. Its use in intractable synovitis and osteoarthritis appears particularly attractive. To date, no randomized controlled study has been conducted to assess the analgesic effects of arterial embolization in patients with symptomatic TKR. A study of 12 patients at the CHU de NICE showed good tolerance of the technique and a significant effect on the KOOS 12 pain score, which improved by 38% at 3 and 6 months. In view of the results of this study, and in this situation of therapeutic impasse, it seems appropriate to evaluate this technique in a randomized, controlled therapeutic trial, which could offer real therapeutic hope

The main objective this double-blind (patient and evaluator), randomized, prospective study is to evaluate the effectiveness of embolization on the pain of patients with persistent pain on a total knee prosthesis by double-blind comparison of two groups at 3-months: the first control group (sham) will include patients who will benefit from arteriography and an injection of saline in their neovessels. The second group, called treatment group, will consist of patients whose neovessels will be occluded by inert microparticles of 100 µm. The pain will be evaluated in both groups before and 3 months after embolisation. The objective is to show that the pain is significantly less important in the group of patients whose neovessels have been occluded with microparticles in comparison to the control group.

Secondary objectives are to evaluate the effectiveness of neovascular embolization on pain, symptoms and functional limitation, knee stiffness, physical activity, quality of life, use of analgesics and anti-inflammatories over the 12 month-follow-up period. The safety and the medico-economic impact will also be evaluated.

Study Population: 112 patients aged 40 to 80 years with a painful total prosthesis with a visual analogue scale (VAS) score greater than or equal to 40 mm for at least 3 months despite an optimal medical treatment, and investigations ruling out malpositioning, loosening and sepsis of the prosthesis,

Primary endpoint: modification of the pain item of the self-administered 12-item Knee injury and Osteoarthritis Outcome Score (KOOS-12) between baseline and 3 months.

Secondary evaluation criteria are KOOS-12, VAS (visual analogic scale), AMIQUAL (Quality of Life Scale) at baseline and then at 6 months; the use of analgesics and anti-inflammatories; adverse effects, medico-economic impact of embolization.

Expected benefits: This study should contribute to improving knowledge in the field of knee prostheses and, more generally, knee osteoarthritis and its management. More importantly, should the study prove conclusive, the results would enable us to extend the use of embolization treatment to all patients with chronic pain following knee prosthesis. At a societal level, health savings could be envisaged thanks to lower consumption of care and prolonged autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged between 40 and 80 years with a TKR for more than one year.
* TKR pain with a VAS ≥ 40 mm having progressed for at least 3 months despite the initiation of a well-conducted medical treatment including stage I and II analgesics and NSAIDs in the absence of contraindication.
* Investigations within 6 months to rule out malposition, loosening and sepsis (conventional X-rays, bone scan, knee CT scan and biological work-up for inflammatory syndrome).
* No revision surgery envisaged.
* Echodoppler hyperemia over the painful area of the knee.
* Subjects affiliated to social security.
* Signed consent to the study.

Exclusion Criteria:

* Local infection of the TKR or systemic infection.
* Algoneurodystrophy.
* Prosthesis loosening.
* Neuropathic pain.
* Allergy to contrast media.
* Fibromyalgia.
* Chronic or acute renal failure (clearance < 30 ml/mn).
* Hemostasis disorders (platelet count < 50,000/mm3 or patient activated partial thromboplastin time (aPTT)/control aPTT>1.2 or prothrombin ratio < 50%).
* Operative indication for removal of the prosthesis retained
* Patient with severe obliterative arteriopathy of the lower limbs (Leriche et Fontaine stage 3).
* Lidocaine contraindication: known hypersensitivity to lidocaine hydrochloride, amide-bonded local anesthetics or any of the excipients; patients with recurrent porphyria.
* Vulnerable persons (minors, patients under guardianship or curatorship, deprived of liberty, under court protection, etc.).
* Pregnant patients: for patients of childbearing age, a pregnancy test will be performed during the screening visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Evolution of the pain assessed by Pain item of the Knee injury and Osteoarthritis Outcome Score 12 (KOOS 12) at 3 months | before intervention and at month 3
  The effectiveness of embolization will be determined by pain assessment using the pain item of the Knee injury and Osteoarthritis Outcome Score 12 (KOOS 12) self-questionnaire (score 0-100). The evolution of this pain score between M0 and M3 will be calculated. KOOS 12 is a self-administered questionnaire that measures patients' perceptions of their knee health, symptoms and functionality. The KOOS-12 comprises 4 items relating to pain, 4 items relating to function (activities of daily living, sport and recreation) and 4 items relating to quality of life.

SECONDARY OUTCOMES:
Evolution of pain throughout the patient's follow-up period assessed by KOOS 12 pain score | From before intervention to Month 12.
  The evolution of pain will be measured here by the KOOS 12 pain score, as in the main objective. The KOOS 12 pain score will be collected at Month 0, Month 1, Month 3, Month 6 and Month 12.
Progression of patient's symptoms and functional limitations throughout the patient's follow-up period assessed by global KOOS score | From before intervention to Month 12.
  The patient's symptoms and functional limitations will be assessed using the global KOOS 12 score (score from 0 to 100). The global KOOS 12 score will be collected at Month 0, Month 1, Month 3, Month 6 and Month 12.
Evolution of pain throughout the patient's follow-up period assessed by VAS (Visual Analog Score) | From before intervention to Month 12.
  Pain will be measured using a VAS (Visual Analog Scale). The VAS will be graduated from 0 to 100 mm, with 0 = no pain and 100 = maximum pain perceived in the 48 hours preceding the consultation, as recommended by the OARSI in osteoarthritis on pain assessment.The pain VAS will be collected at Month 0, Month 1, Month 3, Month 6 and Month 12.
Evolution of Quality of Life throughout the patient's follow-up period, assessed by the AMIQUAL (Arthrose des Membres Inférieurs et QUAlité de vie) Score | From before intervention to Month 12
  Quality of life (QoL) will be measured using the AMIQUAL score. This score is a quality-of-life instrument specific to hip and knee osteoarthritis, capable of capturing patients' perception of their disease.It comprises 5 domains: physical activity (19 items), mental health (14 items), social support (4 items), social functioning (3 items) and pain (3 items), plus 3 items relating to family, sexuality and work. Each item is scored from 1-10, with lower scores reflecting better quality of life. QoL will be collected during patient follow-up at Month 0, Month 3 and Month 12.
Analgesic and anti-inflammatory drugs consumption throughout the the patient's follow-up period | From before intervention to Month 12
  This consumption will be evaluated by the number of days with anti-inflammatory drugs and the number of days with analgesics during the follow-up from Month 0 to Month 6. This information will be collected by the patient in a notebook provided specifically for this purpose. Patients will simply be asked to record the days on which they took anti-inflammatory drugs and analgesics in relation to their knee pain.
Incidence of Serious Adverse Events (safety) throughout the study | From consent signature to Month12
  Adverse events will be recorded throughout the sudy. Safety will be assessed by incidence of Serious Adverse Events.
Medico-economic impact assessed by the incremental cost-effectiveness ratio throughout the study | From before intervention to Month 12
  The medico-economic impact is assessed by the incremental cost-effectiveness ratio in terms of cost per patient with at least a 50% reduction in the KOOS 12 pain score throughout the study.
Medico-economic impact assessed by the incremental cost-utility ratio throughout the study | From before intervention to Month 12
  The medico-economic impact is assessed by the incremental cost-utility ratio in terms of cost per quality-adjusted life year (QALY) gained. The EQ-5D-5L (EuroQol questionnaire 5-Dimensions-5 Levels) comprises a descriptive system and a visual analog scale (VAS). The descriptive system comprises 5 items representing 5 dimensions (mobility, autonomy, daily activities, pain/grief and anxiety/depression) with five levels of health status (no problems, mild problems, moderate problems, severe problems and extreme problems/incapacity). For each of the 5 dimensions, the patient's response is converted into a number between 1 and 5. The 5 numbers obtained are then combined to produce a five-digit score describing the patient's state of health, which is then converted into a utility value (For France : utility value of between -0.53 (health worse than death) and 1 (best possible health). The VAS records the respondent's self-assessed state of health (scale 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Roux, Pr, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (11):
- France (11):
  - Centre Hospitalier Henri Mondor, Créteil
  - Centre Hospitalier Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Saint-Philibert, Lomme
  - Hôpital Saint Philibert, Lomme
  - CHU Marseille, Marseille
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier de Nîmes, Nîmes
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Antoine, Paris
  - Hospices Civils de Strasbourg, Strasbourg